CLINICAL TRIAL: NCT03198143
Title: Effect of Ghrelin on Nutritional and Financial Decision-Making
Brief Title: Effect of Ghrelin on Decision-Making
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: Jenny Tong, MD, MPH (Other)
Responsible Party: Sponsor-Investigator, Jenny Tong, MD, MPH, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00077515
Record Dates: First submitted 2017-05-25; First posted 2017-06-26 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers; Obesity
Keywords: Decision-making; Ghrelin; Healthy Volunteers; Obese
MeSH Terms: conditions — Obesity | interventions — Ghrelin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Subjects - Ghrelin (Experimental): Healthy subjects will arrive after consuming a standard meal 60 minutes prior to study onset. They will receive a single subcutaneous injection of human synthetic Acyl Ghrelin at the start of the study. 5 minutes post-injection, the subjects will receive written instructions and begin their first decision-making task on a computer.
  Interventions: Drug: Ghrelin
- Healthy Subjects - Saline (Placebo Comparator): Healthy subjects will arrive after consuming a standard meal 60 minutes prior to study onset. They will receive a single subcutaneous injection of 0.9% saline at the start of the study. 5 minutes post-injection, the subjects will receive written instructions and begin their first decision-making task on a computer.
  Interventions: Drug: Saline
- Obese Subjects - Ghrelin (Experimental): Obese subjects will arrive after consuming a standard meal 60 minutes prior to study onset. They will receive a single subcutaneous injection of human synthetic Acyl Ghrelin at the start of the study. 5 minutes post-injection, the subjects will receive written instructions and begin their first decision-making task on a computer.
  Interventions: Drug: Ghrelin
- Obese Subjects - Saline (Placebo Comparator): Obese subjects will arrive after consuming a standard meal 60 minutes prior to study onset. They will receive a single subcutaneous injection of 0.9% saline at the start of the study. 5 minutes post-injection, the subjects will receive written instructions and begin their first decision-making task on a computer.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ghrelin — Subjects will receive a subcutaneous injection of synthetic acyl ghrelin (12 µg/kg) at the start of the study.
  Other Names: Acylated Ghrelin; Octanoyl Ghrelin
  Arms: Healthy Subjects - Ghrelin; Obese Subjects - Ghrelin
Drug: Saline — Subjects will receive a subcutaneous injection of saline (0.9%) at the start of the study.
  Arms: Healthy Subjects - Saline; Obese Subjects - Saline

SUMMARY:
This study evaluates the effect of the "hunger hormone" ghrelin on human decision-making. Participants will be given an injection of ghrelin or saline on different study days and will then be asked to make a series of computer-based decisions. The investigators hypothesize that ghrelin will increase participant's preference for energy-dense foods and will also increase impulsiveness in decision making.

DETAILED DESCRIPTION:
Ghrelin is a hormone made by the stomach that stimulates hunger and feeding behavior. How ghrelin affects human decision-making is poorly understood. This study will investigate the effect of ghrelin on nutrition-related and time-based decisions in humans. Participants eye movements will be tracked by a computer during the decision-making process.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and understand English
* BMI of 18.0 - 24.9 kg/m2 or 30.0 - 50.0 kg/m2

Exclusion Criteria:

* Diagnosis of diabetes mellitus (including gestational diabetes)
* Active infections
* History of malignant or inflammatory conditions, such as rheumatoid arthritis and inflammatory bowel disease
* History of myocardial infarction or congestive heart failure
* Active liver or kidney disease
* Uncontrolled hypertension
* Pituitary or adrenal disorders or neuroendocrine tumors
* History of anorexia nervosa, bulimia, or eating disorders not otherwise specified (NOS); Score of "at risk" on the EAT-26 eating disorder screening tool
* Diagnosis of attention-deficient/hyperactivity disorder (ADHD)
* Malabsorptive gastrointestinal disease, gastroparesis, or history of gastrointestinal surgery
* Pregnancy or lactation
* Requirement of daily medications that alter gastrointestinal function (including, but not limited to, glucocorticoids, psychotropics, narcotics, and metoclopramide).
* Requirement of glasses for impaired vision (including reading glasses). Subjects who wear contact lenses for vision correction will not be excluded.
* Insufficient visual acuity to read and interpret the decision stimuli
* Insufficient motor capabilities to press a button, move the joystick, or move their eyes to indicate a response

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Effect of Ghrelin on food choices in Task 1. | Approximately 25 minutes
  The difference in the proportion of healthy and unhealthy choices in the Saline and Ghrelin conditions.
Effect of Ghrelin on temporal choices in Task 2 | Approximately 25 minutes
  The difference in the proportion of smaller sooner and larger later choices in the Saline and Ghrelin conditions

SECONDARY OUTCOMES:
Dwell time on each choice during Task 1 | Approximately 25 minutes
  For eye-tracking, total dwell time (in ms) on each item in a food choice will be compared in both experimental conditions.
Number of fixations on foods during Task 1 | Approximately 25 minutes
  The total number of fixations on each food option will be compared in both experimental conditions.
Dwell time on each choice during Task 2 | Approximately 25 minutes
  For eye-tracking, total dwell time (in ms) on each item in the monetary choice will be compared in both experimental conditions.
Number of fixations on foods during Task 2 | Approximately 25 minutes
  The total number of fixations on each monetary option will be compared in both experimental conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Tong, MD, MPH, Principal Investigator — Duke Molecular Physiology Institute
Locations (1):
- Duke Sociology-Psychology Building 417 Chapel Drive, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No